CLINICAL TRIAL: NCT01418287
Title: An Observational Study to Characterize Children and Adults With Influenza Like Illness (ILI) in Mexico
Brief Title: Characterization of Influenza-like Illness in Mexico
Status: Completed | Type: Observational
Sponsor: Mexican Emerging Infectious Diseases Clinical Research Network (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Secretaria de Salud, Mexico (Other Government); Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other); Instituto Nacional de Enfermedades Respiratorias (Other Government); National Institute of Pediatrics, Mexico (Other Government); Hospital General Dr. Manuel Gea González (Other Government); Hospital Infantil de Mexico Federico Gomez (Other); Hospital Central "Dr. Ignacio Morones Prieto" (Other)
Responsible Party: Sponsor
Other Study IDs: ILI002; HHSN272200900003I (Other Grant/Funding Number: National Institute of Allergy and Infectious Diseases)
Record Dates: First submitted 2011-08-15; First posted 2011-08-17 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Influenza-like Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, PBMC and Nasopharingeal aspirates
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hospitalized: Subjects who are hospitalized due to influenza-like illness
- Non-hospitalized: Subjects who are not hospitalized

SUMMARY:
A study to characterize children and adults with influenza like symptoms and to determine risk factors for severe disease and death among those with H1N1.

DETAILED DESCRIPTION:
In March 2009, a new influenza A virus, novel H1N1 (commonly referred to as "swine flu"), began causing an increase in reports of influenza-like illness in North America. Although the virus subsequently spread rapidly around the world, the earliest reported outbreak of cases occurred in Mexico City, which is seen as the epicenter of the influenza pandemic, the world's first in 40 years.

Many questions remain about this emerging pandemic and the virus causing it, the answers to which could better inform patient management and policy decisions both in Mexico and internationally. Sparse reliable clinical research data have been collected on the natural history of the disease, on the risk factors associated with severe disease, or on the severity of this pandemic influenza as compared to seasonal influenzas. This study is an initial step to better characterize individuals in Mexico who develop influenza-like illness (including illness caused by novel H1N1), to describe the clinical management of those individuals, and to assess their short-term outcome. The planned data collection will provide timely information to inform policy and guidelines for the local populations and governments involved and may also be used to design future ancillary studies of this influenza virus and/or studies of other emerging infectious diseases.

The purpose of this observational study is to characterize individuals in Mexico who seek medical care for influenza-like illness (ILI) and to describe clinical course over a period of at least 28 days after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent by participant, or for pediatric participants, signed informed consent by parent/legal guardian and, where appropriate, signed assent by participant
* At least one respiratory symptom (e.g., shortness of breath, postnasal drip, cough) and
* One of the following criteria:
* Fever (≥ 38 °C by any method: oral, axillary, etc.) on examination or participant-reported fever (≥ 38° C) or feverishness in the past 24 hours
* One or more non-respiratory symptoms (e.g., malaise, headache, myalgia,chest pain)
* Consenting to provide aspirate or naso-pharyngeal swab

Exclusion Criteria

* The onset of illness is more than 48 hours after hospitalization.
* Participants previously included in this study within the last 30 days.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with influenza-like illness presenting to clinical sites in Mexico
Sampling Method: Non-Probability Sample
Enrollment: 5819 (Actual)
Dates: Start 2010-04; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Characterize individuals who develop influenza-like illness, influenza A, and/or H1N1 or other viruses | 5 years
  Characterize demographics, co-morbid conditions, prior influenza vaccination, the use of antivirals, and clinical course and treatment

SECONDARY OUTCOMES:
Death | 5 years
  For all participants, to estimate the percentage who die
Hospitalization | 5 years
  For all participants, to estimate the percentages who require hospitalization due to severe influenza
Risk factors | 5 years
  For all participants, to determine risk factors for severe disease
Repository of oropharyngeal and nasal samples | 5 years
  Establish a repository of oropharyngeal and nasal samples to determine a precise diagnosis, to molecularly characterize the virus
Repository of serum and PBMC | 5 years
  Establish a repository of serum and PBMC to study biomarkers that predispose and correlate with severe influenza

CONTACTS AND LOCATIONS:
Overall Officials: Arturo Galindo Fraga, Dr., Principal Investigator — Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán (INCMNSZ); Ana Alejandra Ortiz Hernández, Dr., Principal Investigator — Instituto Nacional de Pediatría
Locations (6):
- Mexico (6):
  - Instituto Nacional de Pediatría (INP), México, State of Mexico
  - Hospital Infantil de México Federico Gómez (HIM), México, State of Mexico
  - Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán (INCMNSZ), México, State of Mexico
  - Hospital General y de Alta Especialidad Dr. Manuel Gea González, México, State of Mexico
  - Instituto Nacional de Enfermedades Respiratorias (INER), México, State of Mexico
  - San Luis Potosí (SLP):Hospital Central Dr. Ignacio Morones Prieto/Universidad Autónoma de San Luis Potosí, San Luis Potosí City

REFERENCES:
- [Derived] Galindo-Fraga A, Guerra-de-Blas PDC, Ortega-Villa AM, Mateja A, Ruiz Quinones JA, Ramos Cervantes P, Ledesma Barrientos F, Ortiz-Hernandez AA, Llamosas-Gallardo B, Ramirez-Venegas A, Valdez Vazquez R, Noyola Chepitel D, Moreno-Espinosa S, Powers JH, Guerrero ML, Ruiz-Palacios GM, Beigel JH; Mexican Emerging Infectious Diseases Network. Different Clinical Presentations of Human Rhinovirus Species Infection in Children and Adults in Mexico. Open Forum Infect Dis. 2022 Jun 17;9(7):ofac303. doi: 10.1093/ofid/ofac303. eCollection 2022 Jul. PMID 35891697
- [Derived] Galindo-Fraga A, Ortiz-Hernandez AA, Ramirez-Venegas A, Vazquez RV, Moreno-Espinosa S, Llamosas-Gallardo B, Perez-Patrigeon S, Salinger M, Freimanis L, Huang CY, Gu W, Guerrero ML, Beigel J, Ruiz-Palacios GM; La Red ILI 002 Study Group. Clinical characteristics and outcomes of influenza and other influenza-like illnesses in Mexico City. Int J Infect Dis. 2013 Jul;17(7):e510-7. doi: 10.1016/j.ijid.2013.01.006. Epub 2013 Feb 14. PMID 23416208